CLINICAL TRIAL: NCT03453151
Title: Splanchnic Nerve Blockade in Chronic Heart Failure. Splanchnic CHF
Brief Title: Abdominal Nerve Blockade in Chronic Heart Failure.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090299
Record Dates: First submitted 2018-02-20; First posted 2018-03-05 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Regional nerve anesthesia (Experimental)
  Interventions: Drug: splanchnic nerve anesthesia with a local anesthetic

INTERVENTIONS:
Drug: splanchnic nerve anesthesia with a local anesthetic — regional nerve block with a local anesthetic (Lidocaine/Bupivacaine)

SUMMARY:
Patients with chronic heart failure and undergoing right heart catheterization will be enrolled in this study. Subjects will undergo catheterization of the heart to obtain central cardiac pressure and other cardiac hemodynamic parameters. Subsequently, the subject will undergo a regional nerve block of the splanchnic nerves.

This study will be a prospective, uncontrolled clinical trial. The study will not be controlled as invasive monitoring of hemodynamics will be performed, allowing clear demonstration of a cause-effect relationship. The goal of the study is to provide proof of concept.

Patients will undergo detailed physiological testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure (HF)
* Symptomatic with dyspnea
* On a stable HF drug regimen

Exclusion Criteria:

* Ongoing treatment with oral anticoagulation other than aspirin
* Immunosuppressive medications for solid organ transplant
* Acute MI (STEMI or Type I NSTEMI) within 7 days
* Systolic blood pressure < 90 mmHg or >180 mmHg
* Infiltrative cardiomyopathy or constrictive cardiomyopathy
* Chronic kidney disease stage 5
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manesh Patel, Principal Investigator — Duke University
Locations (1):
- Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kittipibul V, Ganesh A, Coburn A, Coyne BJ, Gray JM, Molinger J, Ray N, Podgoreanu M, McCartney SL, Mamoun N, Fitzhugh RC, Lurz P, Green CL, Hernandez AF, Patel MR, Fudim M. Splanchnic Nerve Modulation Effects on Surrogate Measures of Venous Capacitance. J Am Heart Assoc. 2023 Jul 18;12(14):e028780. doi: 10.1161/JAHA.122.028780. Epub 2023 Jul 14. PMID 37449573
- [Derived] Fudim M, Patel MR, Boortz-Marx R, Borlaug BA, DeVore AD, Ganesh A, Green CL, Lopes RD, Mentz RJ, Patel CB, Rogers JG, Felker GM, Hernandez AF, Sunagawa K, Burkhoff D. Splanchnic Nerve Block Mediated Changes in Stressed Blood Volume in Heart Failure. JACC Heart Fail. 2021 Apr;9(4):293-300. doi: 10.1016/j.jchf.2020.12.006. Epub 2021 Mar 10. PMID 33714749
- [Derived] Fudim M, Boortz-Marx RL, Ganesh A, DeVore AD, Patel CB, Rogers JG, Coburn A, Johnson I, Paul A, Coyne BJ, Rao SV, Gutierrez JA, Kiefer TL, Kong DF, Green CL, Jones WS, Felker GM, Hernandez AF, Patel MR. Splanchnic Nerve Block for Chronic Heart Failure. JACC Heart Fail. 2020 Sep;8(9):742-752. doi: 10.1016/j.jchf.2020.04.010. Epub 2020 Jun 10. PMID 32535123

RESULTS

PARTICIPANT FLOW:
Groups:
- Splanchnic Nerve Block (SNB): Splanchnic nerve anesthesia with a local anesthetic: regional nerve block with a local anesthetic (Lidocaine/Ropivacaine)
Period: Overall Study
Arm/Group | Splanchnic Nerve Block (SNB)
Started | 19
Completed | 15
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Participants who completed the study.
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
N terminal pro BNP (B-type natriuretic peptide) level [Mean (Full Range); unit: pmol/L] | 2172 [112 to 9319]

OUTCOME MEASURES:

1. Primary Outcome: Exercise Capacity as Measured by Peak Oxygen Uptake (Peak VO2)
Description: Peak VO2 will be measured before and after nerve block.
Time Frame: baseline, up to 1 hour
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
mL/kg/min
  Before nerve block | 9.1 (2.5)
  After nerve block | 9.8 (2.7)
Statistical Analysis 1: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p = 0.053, Paired t-test

2. Primary Outcome: Mean Pulmonary Arterial Pressure (mPAP)
Description: Mean pulmonary arterial pressure will be measured before and after nerve block.
Time Frame: baseline, up to 1 hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
mmHg
  Before nerve block | 40.5 (12.3)
  After nerve block | 32.7 (13.8)
Statistical Analysis 1: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p < 0.001, Paired t-test

3. Primary Outcome: Pulmonary Capillary Wedge Pressure (PCWP)
Description: Pulmonary capillary wedge pressure will be measured at 20 Watts steady state and peak exercise.
Time Frame: baseline, up to 1 hour
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
mmHg
  Steady state, before nerve block | 28.3 (7.6)
  Steady state, after nerve block | 20.3 (9.5)
  Peak exercise, before nerve block | 34.8 (10.0)
  Peak exercise, after nerve block | 25.1 (10.7)
Statistical Analysis 1: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p < 0.001, Paired t-test

4. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac index will be measured at 20 Watts steady state and peak exercise. Cardiac index (CI) is a haemodynamic parameter that relates the cardiac output (CO) from left ventricle in one minute to body surface area (BSA), thus relating heart performance to the size of the individual.
Time Frame: baseline, up to 1 hour
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
L/min/m^2
  Steady state, before nerve block | 1.9 (0.6)
  Steady state, after nerve block | 2.3 (0.7)
  Peak exercise, before nerve block | 3.4 (1.2)
  Peak exercise, after nerve block | 3.8 (1.1)
Statistical Analysis 1: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p = 0.077, Paired t-test; This analysis refers to the resting cardiac index
Statistical Analysis 2: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p = 0.069, Paired t-test; This analysis refers to the peak exercise cardiac index

5. Secondary Outcome: Urine Output
Description: Urine output will be measured in the 2 hours before the nerve block and in the 2 hours afterwards
Time Frame: 2 hours pre-SNB, 2 hours post-SNB
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
mL
  Before nerve block | 167 (174)
  After nerve block | 297 (180)

6. Secondary Outcome: Renal Biomarker Levels
Description: BUN (blood urea nitrogen) and creatinine levels will be measured in the 2 hours before the nerve block and in the 2 hours afterwards.
Time Frame: 2 hours pre-SNB, 2 hours post-SNB
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Splanchnic Nerve Block (SNB)
Number analyzed (Participants) | 15
mg/dL
  Creatinine, before nerve block | 1.2 (0.4)
  Creatinine, after nerve block | 1.2 (0.4)
  BUN, before nerve block | 19 (10)
  BUN, after nerve block | 18 (10)
Statistical Analysis 1: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p = 0.250, Paired t-test; This analysis refers to creatinine level
Statistical Analysis 2: Comparison: Splanchnic Nerve Block (SNB); Test type: Other; p = 0.014, Paired t-test; This analysis refers to BUN level

ADVERSE EVENTS:
Time Frame: 48 hours after SNB
Groups:
- Splanchnic Nerve Block: Splanchnic nerve anesthesia with a local anesthetic: regional nerve block with a local anesthetic (Lidocaine/Ropivacaine)
Arm/Group | Splanchnic Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Splanchnic Nerve Block (N=15)
Diarrhea (Gastrointestinal disorders) | 1 (1) — Diarrhea for <24 hours
Orthostasis (Cardiac disorders) | 4 (4) — The first five patients had bilateral SNB and four of them developed symptomatic orthostatic hypotension (systolic blood pressure drop >20mmHg with 5 min standing). In all cases the orthostatic hypotension resolved with oral or intravenous hydration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT03453151/Prot_SAP_000.pdf